CLINICAL TRIAL: NCT02879435
Title: Management of Postoperative Pain With Preemptive Analgesia in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mark Kosanovich (Other)
Responsible Party: Sponsor-Investigator, Mark Kosanovich, Doctor, Mercy Hospital and Medical Center, Illinois
Organization: Mercy Hospital and Medical Center, Illinois (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-0401
Record Dates: First submitted 2016-06-17; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine (Experimental): Intervention
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): Control
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupivacaine — pre-operative wound infiltration with 10 ml of numbing medicine
  Other Names: Marcaine
  Arms: bupivacaine
Other: Placebo — pre-operative wound infiltration with 10 ml of sterile water
  Arms: Placebo

SUMMARY:
This research will explore the question of whether preincisional skin infiltration with bupivacaine 0.25% decreases postoperative pain after Cesarean delivery.

DETAILED DESCRIPTION:
Labor and delivery is a time of intense pain, often influenced by the psychological, emotional, social, cultural, and physical state of the parturient. Nowadays, delivery by Cesarean section is becoming more frequent. Females undergoing Cesarean section often wish to be awake postoperatively and to avoid excessive medications that will affect interactions with their newborn infant and visitors. However, Cesarean delivery is often associated with severe pain, requiring a well-planned analgesia regimen to ensure adequate patient comfort and satisfaction, early mobilization, and to decrease the hospital stay. An analgesic regimen may often include multiple doses of IV NSAIDs and opioids to adequately control the pain, and these costs add to the expenses of the hospital stay. Therefore, any intervention that leads to improvement in pain relief is worthy of investigation. Subcutaneous administration of local anesthetics can be a method of postoperative pain control after Cesarean section. Bupivacaine, a widely used local anesthetic, has been studied extensively in the past for the management of postoperative pain. The postoperative analgesic effects of subcutaneous wound infiltration prior to incision with bupivacaine have not been extensively studied in Cesarean delivery; hence, there may be a role in the management of pain relief when bupivacaine is administered at a specific time in surgery. Therefore, the present study is designed to assess the effect of preincisional skin infiltration with bupivacaine 0.25% versus placebo on postoperative pain relief after Cesarean delivery. 120 pregnant patients are randomized by means of the Drug Randomization Protocol (see below). The two groups are (A) control group in which preoperative wound infiltration with 10ml of 0.9% preservative-free normal saline is administered; and (B) in which preoperative wound infiltration with 10ml of 0.25% bupivacaine is administered. The primary end-point is postoperative pain. On arrival to the recovery room, pain intensity at rest is assessed by visual analogous scale ranging from 0 (no pain) to 10 (worst pain imaginable) and then 15, 30, 60 minutes and then 120 minutes after arrival in the recovery room.

Drug Randomization Protocol - All surgical staff is blinded to the study drug contents. A randomization checklist created by the Mercy biostatistician will be given to the scrub technician with a randomly generated list of 1s (saline) and 2s (bupivicaine) indicating the study drug to be administered. The scrub technician will assign a study drug to each patient as they arrive sequentially following the Study Randomization Checklist. The pharmacist will have the master list, indicating the contents of study drug 1 and 2. The scrub technician will order the study drug from the pharmacist by study name and number, eg. "Kathy Tom's study, drug 1." The pharmacist will be instructed not to indicate what the contents of the study related drug to the scrub technician or surgical staff and will send the drug up in a syringe labeled "Kathy Tom Study - Drug #" with all drug descriptive labeling covered.

The Study Randomization Checklist indicates the sequential participant number assigned to the patient on study entry, the corresponding study drug to be administered with a check box to indicate that the drug has been successfully administered (the box will not be checked if ordered and not administered), a column to record the date that the study drug has been administered, a column surgical to record the technician's initials that requested the study drug, and the medical record number of the patient. Sufficient information is included on the checklist to connect the study drug back to the patient if it becomes necessary.

ELIGIBILITY:
Inclusion Criteria:

* adult pregnant women to age 45 with scheduled cesarean sections at Mercy Hospital and Medical Center

Exclusion Criteria:

* Emergent cesarean sections and subjects with contraindications to bupivacaine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Final score on the visual analogous scale | 120 minutes after arrival in the recovery room

SECONDARY OUTCOMES:
Additional amount of analgesia provided patient as part of routine care | Post 120 minutes after arrival in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Rohitkumar Vasa, MD, Study Chair — IRB Chair
Locations (1):
- Mercy Hospital & Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No